CLINICAL TRIAL: NCT02616770
Title: Phase1, Placebo-Controlled, Randomized, Double-blind, Single-ascending Dose Study to Evaluate the Safety and Tolerability of S-1226 Administered by Nebulization in Normal Health Volunteers
Brief Title: Phase1, Placebo-Controlled, Randomized, Double-blind, Single-ascending Dose Study in Healthy Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SolAeroMed Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: SAMi-01-1-01
Record Dates: First submitted 2015-11-25; First posted 2015-11-30 (Estimated); Last update posted 2015-11-30 (Estimated); Status verified 2014-09

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — perfluorooctylbromide and CO2 drug combination; perflubron; Carbon Dioxide; Sodium Chloride; Air

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- S1226 (4%) (Experimental): S1226 (4%) dosed as single dose for 2 minutes
  Interventions: Drug: S1226 (4%)
- Saline (for 4%) (Placebo Comparator): 3 mL saline and medical air as single dose for 2 minutes
  Interventions: Drug: Saline (for 4%)
- S1226 (8%) (Experimental): S1226 (8%) dosed as single dose for 2 minutes
  Interventions: Drug: S1226(8%)
- Saline (for 8 %) (Placebo Comparator): 3 mL saline and medical air as single dose for 2 minutes
  Interventions: Drug: Saline (for 8%)
- S1226 (12%) (Experimental): S1226 (12%) dosed as single dose for 2 minutes
  Interventions: Drug: S1226(12%)
- Saline (for 12%) (Placebo Comparator): 3 mL saline and medical air as single dose
  Interventions: Drug: Saline (for 12%)

INTERVENTIONS:
Drug: S1226 (4%) — 3 ml Peflubron nebulized, with Medical Gas containing 4% carbon Dioxide, for 2 minutes as a single dose.
  Other Names: Perflubron and Medical Gas containing 4% Carbon Dioxide
  Arms: S1226 (4%)
Drug: Saline (for 4%) — 3ml saline nebulized, with Medical Air, for 2 minutes as a single dose
  Other Names: Saline and Medical Air
  Arms: Saline (for 4%)
Drug: S1226(8%) — 3 ml Peflubron nebulized, with Medical Gas containing 8% carbon Dioxide for, 2 minutes as a single dose.
  Other Names: Perflubron and Medical Gas containing 8% Carbon Dioxide
  Arms: S1226 (8%)
Drug: Saline (for 8%) — 3ml saline nebulized, with Medical Air, for 2 minutes as a single dose
  Other Names: Saline and Medical Air
  Arms: Saline (for 8 %)
Drug: S1226(12%) — 3 ml Peflubron nebulized, with Medical Gas containing 12% carbon Dioxide, for 2 minutes as a single dose.
  Other Names: Perflubron and Medical Gas containing 12% Carbon Dioxide
  Arms: S1226 (12%)
Drug: Saline (for 12%) — 3ml saline nebulized with Medical Air for 2 minutes as a single dose
  Other Names: Saline and Medical Air
  Arms: Saline (for 12%)

SUMMARY:
To evaluate the safety and tolerability of S-1226 composed of perflubron with ascending doses of carbon dioxide (4%, 8%, and 12% CO2) administered over 2 minute nebulisation to healthy subjects.

DETAILED DESCRIPTION:
There will be up to 3 cohorts (1 cohort per dose level). Each cohort will include 12 subjects (9 receiving S-1226 and 3 receiving matching placebo). For each dose level, a sentinel group of 2 subjects will be dosed (1 subject with S-1226, 1 subject with placebo) 24 hours prior to dosing the rest of the study population.

It may be necessary to repeat, or modify (decrease) a dose level, and thus an additional cohort of up to 12 subjects may be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, non-smoker, ≥18 and ≤55 years of age with BMI > 18.5 and < 30.0.
2. Healthy as defined by:

   * the absence of clinically significant illness and surgery within 4 weeks prior to dosing. Subjects vomiting within 24 hours pre-dose will be carefully evaluated for upcoming illness/disease. Inclusion pre-dosing is at the discretion of the Qualified Investigator;
   * the absence of clinically significant history of neurological, endocrinal, cardiovascular, pulmonary, hematological, immunologic, psychiatric, gastrointestinal, renal, hepatic, and metabolic disease;
   * the absence of clinically significant respiratory infection in the preceding 6 weeks;
   * the absence of history of malignancy within the past five years, with the exception of successfully treated non-metastatic basal cell or squamous cell carcinomas of the skin and/or localized carcinoma in situ of the cervix;
   * the absence of clinically significant findings on a chest X-Ray at screening.
3. Steroid-naive (i.e. volunteers who are not currently on topical or systemic corticosteroids or those who have not taken any oral or injectable corticosteroid within 60 days prior to study drug administration or have not used any inhaled/ophthalmic/nasal corticosteroid within 30 days prior to study drug administration).
4. Females of childbearing potential who are sexually active with male partner must be willing to use one of the following acceptable contraceptive methods throughout the study and for 30 days after:

   * simultaneous use of intra-uterine contraceptive device without hormone release system placed at least 4 weeks prior to study drug administration, and for the male partner, condom;
   * simultaneous use of diaphragm and for the male partner, male condom and spermicide starting at least 14 days prior to study drug administration;
   * simultaneous use of female condom starting at least 14 days prior to study drug administration, and for the male partner, condom and spermicide;
   * sterile male partner (vasectomized since at least 6 months).
5. Males subjects who are not vasectomized for more than 6 months, and who are sexually active with non-sterile female partner must be willing to use one of the following acceptable contraceptive methods throughout the study and for 30 days after:

   * simultaneous use of condom, and for the female partner, oral contraceptive, or intra-uterine contraceptive device placed at least 4 weeks prior to study drug administration;
   * simultaneous use of male condom, and for the female partner, diaphragm and spermicide ;
   * simultaneous use of male condom, and for the female partner, female condom and spermicide ;
   * Sterile female partners include post-menopausal women (absence of menses for 12 months prior to drug administration) or women who have had a tubal ligation, hysterectomy, or bilateral oophorectomy (at least 6 months prior to drug administration).
6. Capable of consent.
7. Subjects must have a normal lung function (FEV1 ≥ 80 % of predicted and FEV1/FVC > 70 %).

Exclusion Criteria:

1. Any clinically significant abnormality or abnormal laboratory test results found during medical screening or positive test for hepatitis B, hepatitis C, or HIV found during medical screening.
2. Positive urine drug screen or urine cotinine test at screening.
3. Current cigarette smokers or former smokers with a smoking history of greater than 5 pack years or who stopped smoking within the 2 years preceding enrolment in the study. For the determination of pack years, a pack of cigarettes is assumed to contain 20 cigarettes.
4. History of significant allergic reactions (e.g. angioedema, anaphylactic reactions).
5. History of panic disorder or panic attacks
6. Positive pregnancy test at screening.
7. Any reason which, in the opinion of the Investigator (or delegate), would prevent the subject from participating in the study.
8. Clinically significant electrocardiogram (ECG) abnormalities or vital sign abnormalities (systolic blood pressure lower than 90 or over 140 mmHg, diastolic blood pressure lower than 50 or over 90 mmHg, or heart rate less than 50 or over 100 bpm) at screening.
9. History of significant alcohol abuse within one year prior to screening or regular use of alcohol within six months prior to the screening visit (more than fourteen units of alcohol per week [1 Unit = 150 mL of wine, 360 mL of beer, or 45 mL of 40% alcohol]) or positive alcohol breath test at screening.
10. History of significant drug abuse within one year prior to screening or use of soft drugs (such as marijuana) within 3 months prior to the screening visit or hard drugs (such as cocaine, phencyclidine [PCP], and crack) within 1 year prior to screening.
11. Use of an investigational drug within 30 days (90 days for biologics) or participation in an investigational study within 30 days prior to dosing.
12. Use of anticoagulants, immunosuppressives, regular use of non-steroidal anti-inflammatory drugs, use of anti-IgE medication, or any allergen specific immunotherapy within the last 60 days.
13. Use of medication other than non-steroidal topical products without significant systemic absorption:

    * prescription medication (other than the ones listed previously) within 14 days prior to the first dosing;
    * over-the-counter products including natural health products (e.g. food supplements and herbal supplements) within 7 days prior to the first dosing, with the exception of the occasional use of acetaminophen (up to 2 g daily);
    * a depot injection or an implant of any drug within 3 months prior to the first dosing.
    * monoamine oxidase (MAO) inhibitors within 30 days prior to the first dosing.
14. Donation of blood within 7 days prior to dosing. Donation or loss of blood (excluding volume drawn at screening) of 50 mL to 499 mL of blood within 30 days, or more than 499 mL within 56 days prior to dosing.
15. Hemoglobin <128 g/L (males) and <115 g/L (females) and hematocrit <0.37 L/L (males) and <0.32 L/L (females) at screening.
16. Breast-feeding subject.
17. History of wheezing after exercise
18. History of or previous medical diagnosis of asthma

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2014-03; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability to S-1226 assessment by evaluating adverse events, vital signs, 12-lead ECG, clinical laboratory parameters, and physical examination. | 24 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Latifa Yamlahi, MSc, Study Director — Pharma Medica Research, Inc.

REFERENCES:
- [Derived] Green FH, Leigh R, Fadayomi M, Lalli G, Chiu A, Shrestha G, ElShahat SG, Nelson DE, El Mays TY, Pieron CA, Dennis JH. A phase I, placebo-controlled, randomized, double-blind, single ascending dose-ranging study to evaluate the safety and tolerability of a novel biophysical bronchodilator (S-1226) administered by nebulization in healthy volunteers. Trials. 2016 Jul 28;17:361. doi: 10.1186/s13063-016-1489-8. PMID 27464582